CLINICAL TRIAL: NCT00998244
Title: A Randomized, Double-Blind Crossover Study to Evaluate the Effect of a Very Low Carbohydrate Diet on Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Effect of a Very Low Carbohydrate Diet on Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Nicholas Shaheen, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-0623
Record Dates: First submitted 2009-10-02; First posted 2009-10-20 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Gastroesophageal Reflux Disease; Overweight; Acid Reflux Disease
Keywords: low carbohydrate; low fat; diet; overweight; GERD; gastroesophageal reflux disease; acid reflux; heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Overweight; Heartburn | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Very Low Carbohydrate Diet (Experimental): Very Low Carbohydrate Diet
  Interventions: Other: Diet - very low carb or low fat
- Low Fat Diet (Active Comparator): Low Fat Diet
  Interventions: Other: Diet - very low carb or low fat

INTERVENTIONS:
Other: Diet - very low carb or low fat — Diet comparison in Gastroesophageal Reflux Disease

SUMMARY:
The purpose of this research study is to learn if a very low carbohydrate (sugar) diet or traditional low fat diet is able to reduce symptoms related to gastroesophageal reflux disease (GERD) in people who are overweight. Patients with GERD may experience all or some of the following symptoms: stomach acid or partially digested food re-entering the esophagus (which is sometimes referred to as heartburn or regurgitation) and belching. In this study, the investigators also hope to find out if acid in the esophagus is reduced more by a low carbohydrate diet than a low fat diet.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* BMI between 30 kg/m2 and 45 kg/m2

Exclusion Criteria:

* Known history of Barrett's esophagus or esophageal adenocarcinoma
* Previous surgical anti-reflux procedure
* Previous weight loss surgery, including gastric bypass
* Diabetes
* Pregnancy
* Heart Disease
* Unwillingness to discontinue use of proton pump inhibitors (PPI's) or H2-receptor antagonists per study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in distal esophageal acid exposure after initiating a very low carbohydrate diet compared to the decrease seen after initiating a low fat diet | Baseline, 10 days after baseline, and at 25 days after baseline.

SECONDARY OUTCOMES:
The change in serum levels of pro-inflammatory cytokines after initiating a very low carbohydrate diet compared to a traditional low fat diet as measured with blood samples. | Baseline, 10 days after baseline, and at 25 days after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Shaheen, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States